CLINICAL TRIAL: NCT03789474
Title: Impact of Intra-operative Use of Peristaltic Pneumatic Compression Device on Haemodynamics Vis-à-vis Fluid Requirement During General Anaesthesia and Surgery:A Randomized Prospective Study
Brief Title: Does Fluid Requirement Decrease With the Use of Pneumatic Compression Device on Lower Limbs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Rishikesh (Other Government)
Responsible Party: Principal Investigator, Dr. Masaipeta Kesari, Junior resident,Principal Investigator,Department of Anaesthesiology, All India institute of Medical Sciences, Rishikesh., All India Institute of Medical Sciences, Rishikesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AIIMSRishikesh
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Results first posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Fluid Overload
MeSH Terms: conditions — Edema

STUDY DESIGN:
Intervention Model Description: About 60 patients of age group 25 to 50 belonging to American Society of Anesthesiologists (ASA) grade 1 and 2 were allocated to either control or sequential pneumatic compression device group .Allocation was done by sealed envelop technique.In the operating room,in the control group,the device was placed on operating table and was placed next to the patients calves.in the intervention group,the device was placed over calves and inflated during induction of General Anaesthesia (GA) and maintenance.legs were draped in both the groups.Femoral vein velocities were assessed using ultrasound in preoperative period , intraoperatively 15 minutes after induction of anaesthesia and in post-operative period.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Draping of the legs was done in both the groups.the care observer nor investigator were blinded for the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (No Intervention): No intervention was done ,served as a control group.
- Group B (Experimental): Intervention:peristaltic pneumatic compression device was placed on the legs of the patient and was active. HUNTLEIGH FLOWTRON ACS900 calf length device was used.
  Interventions: Device: HUNTLEIGH FLOWTRON ACS900

INTERVENTIONS:
Device: HUNTLEIGH FLOWTRON ACS900
  Arms: Group B

SUMMARY:
Impact of intraoperative use of pneumatic peristaltic compression device on hemodynamics vis a vis on fluid requirement during general anaesthesia and surgery.

DETAILED DESCRIPTION:
Induction of general anaesthesia is associated with cardiac depression and peripheral vasodilatation resulting in hypotension .This hypotension can be corrected by giving intravenous fluid, or the vasoconstrictor. While optimum fluid balances in the perioperative period is of vital importance in overnight fasting patients to correct the fluid deficit, any fluid overload is not only counterproductive to the heart function but is associated with fluid retention in body and edema in postoperative period.

Peristaltic pneumatic compression device, a variant of intermittent sequential compression of legs, uses higher pressure and longer compression cycles to avoid venous stasis in immobilized patients. Sequential compression devices have sleeves with pockets of inflation, which works to squeeze on the appendage in a milking action .The most distal areas will inflate initially, and the subsequent pockets will follow in the same manner. The primary aim of the device is to squeeze blood from the underlying deep veins to proximal side. When the inflatable sleeves deflate, the veins will replenish with blood. The intermittent compressions of the sleeves will ensure the movement of venous blood . Peristaltic Pneumatic Compression of the legs significantly reduces fluid demand and enhances stability during minor ear, nose, and throat surgery. Peristaltic Pneumatic Compression has the potential to support fluid restriction regimens during surgery .

ELIGIBILITY:
Inclusion Criteria:

* ASA(American Society of Anaesthesiologists) grade I or II, of both genders
* Age group of 25 to 50 years
* Patients undergoing surgeries under GA(General Anaesthesia) for 2-3 hours

Exclusion Criteria:

* Patients expected to get major blood loss
* Burns patients.
* Patients with significant cardiac diseases.
* Patients with pulmonary diseases and impaired renal function.
* Lower limb surgeries and abdominal surgeries

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh Tripathi, MD, Principal Investigator — All India Institute of Medical Sciences, Rishikesh

IPD SHARING:
Plan to Share IPD: Yes
study protocol,stastical analysis plan,informed consent form.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: june 2020 till june 2021
Access Criteria: after obtaining consent.

REFERENCES:
- [Result] Kiefer N, Theis J, Putensen-Himmer G, Hoeft A, Zenker S. Peristaltic pneumatic compression of the legs reduces fluid demand and improves hemodynamic stability during surgery: a randomized, prospective study. Anesthesiology. 2011 Mar;114(3):536-44. doi: 10.1097/ALN.0b013e31820c3973. PMID 21307764
- [Result] Kaufmann KB, Stein L, Bogatyreva L, Ulbrich F, Kaifi JT, Hauschke D, Loop T, Goebel U. Oesophageal Doppler guided goal-directed haemodynamic therapy in thoracic surgery - a single centre randomized parallel-arm trial. Br J Anaesth. 2017 Jun 1;118(6):852-861. doi: 10.1093/bja/aew447. PMID 28575331
- [Result] Meng L, Heerdt PM. Perioperative goal-directed haemodynamic therapy based on flow parameters: a concept in evolution. Br J Anaesth. 2016 Dec;117(suppl 3):iii3-iii17. doi: 10.1093/bja/aew363. PMID 27940452
- [Result] Millard JA, Hill BB, Cook PS, Fenoglio ME, Stahlgren LH. Intermittent sequential pneumatic compression in prevention of venous stasis associated with pneumoperitoneum during laparoscopic cholecystectomy. Arch Surg. 1993 Aug;128(8):914-8; discussion 918-9. doi: 10.1001/archsurg.1993.01420200088016. PMID 8343064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from January 2017 to July 2018 at ALL INDIA INSTITUTE OF MEDICAL SCIENCES,RISHIKESH,UTTARAKHAND ,INDIA.
Groups:
- Group B: Intervention:peristaltic pneumatic compression device was placed on the legs of the patient and was active. HUNTLEIGH FLOWTRON ACS900 calf length device was used.
  HUNTLEIGH FLOWTRON ACS900
Period: Overall Study
Arm/Group | Group A | Group B
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (9.4) | 34.1 (7.6) | 35.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 11 | 12 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: meters] — in meters
  meters | 1.62 (.1) | 1.59 (.1) | 1.60 (.1)
Weight [Mean (Standard Deviation); unit: kilograms] — in kilograms
  kilograms | 60.77 (8.73) | 62.13 (9.1) | 61.45 (8.91)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg^m2] | 22.8 (3.74) | 24.5 (4.2) | 23.65 (3.97)

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate at T0
Description: heart rate monitoring at T0
Time Frame: 15 minutes pre induction
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
beats per minute | 85.23 (17.81) | 88.833 (18.28)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .443, t-test, 2 sided

2. Primary Outcome: Heart Rate at T1
Description: heart rate monitoring at T1
Time Frame: post induction heart rate
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
beats per minute | 79.60 (16.44) | 88.13 (18.35)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .063, t-test, 2 sided

3. Primary Outcome: Heart Rate at T2
Description: heart rate monitoring at T2
Time Frame: 15 minutes after induction
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
beats per minute | 79.97 (13.26) | 88.57 (20.30)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .057, t-test, 2 sided

4. Primary Outcome: Heart Rate at T3
Description: heart rate monitoring at T3
Time Frame: 30 minutes after induction
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
beats per minute | 76.70 (12.26) | 84.77 (16.80)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .038, t-test, 2 sided

5. Primary Outcome: Heart Rate at T4
Description: heart rate monitoring at T4
Time Frame: 60 minutes after induction
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
beats per minute | 77.40 (10.93) | 83.56 (14.83)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .072, t-test, 2 sided

6. Primary Outcome: Heart Rate at T5
Description: heart rate monitoring at T5
Time Frame: 120 minutes after induction
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
beats per minute | 77.53 (12.71) | 82.17 (14.22)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .189, t-test, 2 sided

7. Primary Outcome: Heart Rate at T6
Description: heart rate monitoring at T6
Time Frame: post operative period after 30 min in post anaesthesia care unit
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
beats per minute | 85.06 (12.58) | 88.23 (13.87)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .358, t-test, 2 sided

8. Primary Outcome: Systolic Blood Pressure at T0
Description: systolic blood pressure measurement at T0
Time Frame: 15 min before induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 119.06 (11.71) | 122.1 (16.01)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .406, t-test, 2 sided

9. Primary Outcome: Systolic Blood Pressure at T1
Description: systolic blood pressure measurement at T1
Time Frame: post induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 102.33 (15.31) | 106.80 (14.82)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .256, t-test, 2 sided

10. Primary Outcome: Systolic Blood Pressure at T2
Description: systolic blood pressure measurement at T2
Time Frame: 15 min after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 100.73 (12.12) | 106.93 (13.45)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .066, t-test, 2 sided

11. Primary Outcome: Systolic Blood Pressure at T3
Description: systolic blood pressure measurement at T3
Time Frame: 30 min after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 106.23 (15.08) | 109.90 (12.93)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .316, t-test, 2 sided

12. Primary Outcome: Systolic Blood Pressure at T4
Description: systolic blood pressure measurement at T4
Time Frame: 60 min after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 111.10 (15.59) | 111.23 (12.45)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .971, t-test, 2 sided

13. Primary Outcome: Systolic Blood Pressure at T5
Description: systolic blood pressure measurement at T5
Time Frame: 120 min after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 108.86 (10.92) | 115.70 (12.79)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .030, t-test, 2 sided

14. Primary Outcome: Systolic Blood Pressure at T6
Description: systolic blood pressure measurement at T6
Time Frame: post operative period 30 min in post asnaesthesia care unit
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 118.80 (10.34) | 126.03 (10.49)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .009, t-test, 2 sided

15. Primary Outcome: Diastolic Blood Presure at T0
Description: Diastolic blood pressure measurement at T0
Time Frame: 15 minutes before induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 76.00 (11.66) | 72.23 (13.30)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .704, t-test, 2 sided

16. Primary Outcome: Diastolic Blood Pressure at T1
Description: Diastolic blood pressure measurement at T1
Time Frame: immediately after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 66.30 (12.93) | 69.33 (11.96)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .350, t-test, 2 sided

17. Primary Outcome: Diastolic Blood Pressure at T2
Description: Diastolic blood pressure measurement at T2
Time Frame: 15 minutes after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 65.37 (11.66) | 66.53 (12.29)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .708, t-test, 2 sided

18. Primary Outcome: Diastolic Blood Pressure at T3
Description: Diastolic blood pressure measurement at T3
Time Frame: 30 minutes after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 69.46 (15.42) | 68.13 (12.15)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .711, t-test, 2 sided

19. Primary Outcome: Diastolic Blood Pressure at T4
Description: Diastolic blood pressure measurement at T4
Time Frame: 60 minutes after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 69.36 (16.75) | 69.16 (10.56)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .956, t-test, 2 sided

20. Primary Outcome: Diastolic Blood Pressure at T5
Description: Diastolic blood pressure measurement at T5
Time Frame: 120 minutes after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 66.63 (11.53) | 70.80 (9.93)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .139, t-test, 2 sided

21. Primary Outcome: Diastolic Blood Pressure at T6
Description: Diastolic blood pressure measurement at T6
Time Frame: post induction 30 min in post anaesthesia care unit
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 70.66 (9.80) | 75.80 (8.58)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .035, t-test, 2 sided

22. Primary Outcome: Mean Blood Pressure at T0
Description: Mean blood pressure measurement at T0
Time Frame: 15 minutes pre induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 90.04 (11.03) | 92.19 (13.43)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .502, t-test, 2 sided

23. Primary Outcome: Mean Blood Pressure at T1
Description: Mean blood pressure measurement at T1
Time Frame: immediately after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 78.38 (13.29) | 81.82 (11.89)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .350, t-test, 2 sided

24. Primary Outcome: Mean Blood Pressure at T2
Description: Mean blood pressure measurement at T2
Time Frame: 15 minutes after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 77.38 (11.46) | 79.99 (11.41)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .380, t-test, 2 sided

25. Primary Outcome: Mean Blood Pressure at T3
Description: Mean blood pressure measurement at T3
Time Frame: 30 minutes after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 82.42 (14.36) | 82.05 (11.57)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .914, t-test, 2 sided

26. Primary Outcome: Mean Blood Pressure at T4
Description: Mean blood pressure measurement at T4
Time Frame: 60 minutes after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 83.55 (15.79) | 83.19 (10.14)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .915, t-test, 2 sided

27. Primary Outcome: Mean Blood Pressure at T5
Description: Mean blood pressure measurement at T5
Time Frame: 120 minutes after induction
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 81.16 (10.64) | 85.76 (9.78)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .087, t-test, 2 sided

28. Primary Outcome: Mean Blood Pressure at T6
Description: Mean blood pressure measurement at T6
Time Frame: post operative 30 min in post anaesthesia care unit
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
millimeters of mercury | 86.71 (8.98) | 92.54 (8.27)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .011, t-test, 2 sided

29. Primary Outcome: Femoral Vein Velocity at T0
Description: Femoral vein velocity measuement at T0
Time Frame: 15 minutes pre induction
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters per second | 29.35 (4.20) | 31.31 (7.28)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .207, t-test, 2 sided

30. Primary Outcome: Femoral Vein Velocity at T2
Description: Femoral vein velocity measurement at T2
Time Frame: 15 minutes after induction
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters per second | 27.79 (4.02) | 33.61 (7.61)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .142, t-test, 2 sided

31. Primary Outcome: Femoral Vein Velocity at T6
Description: Femoral vein velocity measurement at T6
Time Frame: after 30 minutes in post anaesthesia care unit
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters per second | 28.35 (5.64) | 31.92 (5.96)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .021, t-test, 2 sided

32. Primary Outcome: Femoral Vein Velocity Variance
Description: the variance in femoral vein velocity was calculated by subtracting the femoral vein velocity pre induction from femoral vein velocity 15 min after induction divided by mean of the two values in percentage
Time Frame: 15 minutes pre induction to 30 minutes in post anaesthesia care unit
Measure: Mean (Standard Deviation); unit: percentage of velocity
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
percentage of velocity | -5.419 (8.444) | 7.188 (5.385)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = 0.0001, t-test, 2 sided

33. Primary Outcome: Femoral Artery Velocity at T0
Description: Femoral artery velocity measurement at T0
Time Frame: 15 minutes pre induction
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters per second | 69.15 (14.08) | 76.25 (13.39)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .030, t-test, 2 sided

34. Primary Outcome: Femoral Artery Velocity at T2
Description: Femoral artery velocity measurement at T2
Time Frame: 15 minutes after induction
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters per second | 67.74 (11.96) | 73.91 (11.62)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .048, t-test, 2 sided

35. Primary Outcome: Femoral Artery Velocity at T6
Description: Femoral artery velocity measurement at T6
Time Frame: after 30 minutes in post anaesthesia care unit
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters per second | 69.82 (11.78) | 76.63 (14.07)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .047, t-test, 2 sided

36. Primary Outcome: Inferior Venacava Diameter (Maximum) at T0
Description: inferior venacava diameter (maximum) meaurement at T0
Time Frame: 15 min pre induction
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters | 1.16 (0.14) | 1.26 (0.17)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .019, t-test, 2 sided

37. Primary Outcome: Inferior Venacava Diameter (Maximum) at T2
Description: inferior venacava diameter (maximum) meaurement at T2
Time Frame: 15 min after induction
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters | 1.27 (0.11) | 1.27 (0.17)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .000, t-test, 2 sided

38. Primary Outcome: Inferior Venacava Diameter (Maximum) at T6
Description: inferior venacava diameter (maximum) meaurement at T6
Time Frame: after 30 min in post anaesthesia care unit
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters | 1.19 (0.13) | 1.31 (0.17)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .004, t-test, 2 sided

39. Primary Outcome: Inferior Venacava Diameter (Minimum) at T0
Description: inferior venacava diameter (minimum) meaurement at T0
Time Frame: 15 min pre induction
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters | 1.06 (0.13) | 1.15 (0.15)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .020, t-test, 2 sided

40. Primary Outcome: Inferior Venacava Diameter (Minimum) at T2
Description: inferior venacava diameter (minimum) meaurement at T2
Time Frame: 15 min after induction
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters | 1.02 (0.09) | 1.15 (0.15)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .000, t-test, 2 sided

41. Primary Outcome: Inferior Venacava Diameter (Minimum) at T6
Description: inferior venacava diameter (minimum) meaurement at T6
Time Frame: after 30 min in post anaesthesia care unit
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
centimeters | 1.11 (0.13) | 1.18 (0.17)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .053, t-test, 2 sided

42. Primary Outcome: Inferior Venacava Diameter Collapsibility Index at T0
Description: the collapsibility index was calculated by dividing the difference of maximum inferior vena cava diameter and minimum inferior vena cava diameter by mean of the two diameters multiplied by 100.This was done for pre induction spontaneously breathing patients
Time Frame: 15 min pre induction
Measure: Mean (Standard Deviation); unit: percentage of diameter
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
percentage of diameter | 9.06 (4.17) | 9.32 (1.62)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .746, t-test, 2 sided

43. Primary Outcome: Inferior Venacava Diameter Distensibility Index at T2
Description: the inferior venacava distensibility index for post induction mechanically ventilated patients. It was calculated by dividing the difference of maximum inferior vena cava diameter and minimum inferior vena cava diameter by minimum inferior vena cava diameters multiplied by 100 .
Time Frame: 15 min after induction
Measure: Mean (Standard Deviation); unit: percentage of diameter
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
percentage of diameter | 11.05 (4.17) | 8.39 (2.841)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .006, t-test, 2 sided

44. Primary Outcome: Inferior Venacava Diameter Collapsibility Index at T6
Description: as for outcome 42
Time Frame: after 30 minutes in post anaesthesia care unit
Measure: Mean (Standard Deviation); unit: percentage of diameter
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
percentage of diameter | 7.04 (3.46) | 10.03 (4.10)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .003, t-test, 2 sided

45. Primary Outcome: FLUID REQUIREMENT (Cumulative)
Description: fluid requirement (cumulative) during the operative period.
Time Frame: operative period
Population: the population is same as the assigned population.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
milliliters | 1456.67 (307.87) | 1291.66 (320.04)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = 0.043, t-test, 2 sided

46. Primary Outcome: Blood Loss During Operation
Description: Total blood loss during operation
Time Frame: During operating procedure
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Group A | Group B
Number analyzed (Participants) | 30 | 30
milliliters | 99.67 (50.34) | 116.67 (41.80)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = .160, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Pre induction to post anaesthesia care unit.
Description: No serious adverse events were reported. No mortality by all cause is reported. No risk for other(not including serious) adverse events is reported.
Groups:
- Group 1: In Group 1 - The PPC was placed on operating table, next to patients calves during the procedure.
- Group 2: In Group 2 - The PPC was placed over calves and inflated during induction of General Anaesthesia and maintenance.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
* Outcome of the patients was not studied.
* The patients studied underwent procedures for short duration of 2-3 hours. Longer procedures were not taken into consideration and the applicability and efficacy in those procedures was not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT03789474/Prot_SAP_ICF_000.pdf